CLINICAL TRIAL: NCT03925415
Title: A National, Observational, Cross-Sectional, Multicenter Study to Estimate the Prevalence of an Eosinophilic Phenotype Among Severe Asthma Patients in Brazil
Brief Title: BRazilian Asthmatics Patients EOSinophilic Profile (BRAEOS)
Acronym: BRAEOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Medical Writer: Dr. Rodrigo Athanazio (Unknown); CRO: CTI-Eurotrials (Unknown)
Responsible Party: Sponsor
Other Study IDs: D3250R00045
Record Dates: First submitted 2019-02-19; First posted 2019-04-24 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Severe Asthma
Keywords: Severe Asthma; Eosinophilic Asthma; Eosinophilic Phenotype
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is a complex and heterogeneous disease. Severe asthma is recognised as a major unmet need that poses a great burden on the healthcare system. While accounting for only a small proportion of the total asthmatic population, asthma-related costs are 1.7 to 4-fold higher than those observed in the mild-persistent asthma population and the associated personal and societal impact is significant.

Severe asthma is not considered to be a single disease, but can be divided into several phenotypes, owing to the variety of inflammatory, clinical and functional characteristics that it can present with. One of the proposed and most studied phenotypes is severe eosinophilic asthma. Patients with severe asthma that is accompanied with a high concentration of eosinophils require greater healthcare resource use, overall greater disease management costs and have a much more impaired QoL than those who do not present with raised eosinophilia.

While the number of targeted treatments for asthma management has been growing in recent years, the heterogeneity of clinical presentations, treatment responses and inflammatory processes involved represents an added challenge for health care professionals. Thus, severe asthma management is a complex endeavour and a thorough and up to date understanding of the pathophysiologic characteristics of the patient population promotes effective therapeutic decision-making.

The purpose of this observational, cross-sectional, multicentre study is to determine the prevalence of an eosinophilic phenotype of blood eosinophil count > 300 cells/mm3 among severe asthma patients followed at Brazilian sites specialized in the management of severe asthma. The prevalence of an atopic phenotype, asthma control, QoL and burden of disease will also be studied.

DETAILED DESCRIPTION:
Knowledge of the prevalence of eosinophilia among adult, severe asthma patients in Brazil is limited. Moreover, data on the prevalence of an atopic phenotype within the adult, severe asthma population is scarce. Severe asthma management is a complex endeavour and a thorough and up to date understanding of the pathophysiologic characteristics of the patient population facilitates therapeutic decisions that effectively lead to disease control.

The purpose of this observational, cross-sectional, multicentre study is to determine the prevalence of an eosinophilic phenotype of blood eosinophil count > 300 cells/mm3 among severe asthma patients followed at Brazilian sites specialized in the management of severe asthma. The prevalence of an atopic phenotype, asthma control, QoL and burden of disease will also be studied. It is expected that this study will contribute to the understanding of severe asthma in Brazil, ultimately helping to inform therapeutic decisions and addressing patients' needs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, aged 18 years or older at the time of study entry.
* Subject followed at a participating centre and attending a routine clinical appointment.
* Subjects with evidence of asthma of either:

  * Documented airway reversibility (forced expiratory volume in one second (FEV1) ≥12% and 200 mL) using the maximum post-bronchodilator procedure OR
  * Documented airway hyperresponsiveness (provocative concentration of methacholine causing a ≥20% fall in FEV1) OR
  * Documented airflow variability in FEV1 ≥20% between two consecutive lung function assessments prior to study entry (FEV1 values recorded during exacerbations should not be considered for this criterion)
* Subjects with a diagnosis of severe asthma for at least one year, according to the criteria of the International ERS/ATS Guidelines on Definition, Evaluation and Treatment of Severe Asthma (6), i.e.:

  * Asthma which requires treatment with guidelines suggested medications for GINA steps 4-5 asthma (high dose ICS (Appendix A) and LABA or leukotriene modifier/theophylline) for the previous year; or
  * Systemic CS for ≥50% of the previous year to prevent it from becoming "uncontrolled" or which remains "uncontrolled" despite this therapy.
* Subject with accurate and complete medical records at the centre.
* Subject that voluntarily signed and dated the informed consent form prior to study entry.

Exclusion Criteria:

* Subjects experiencing a moderate or severe asthma exacerbation as per the Official ATS/ERS Statement on Asthma Control (22) at the time of the study entry, or who had a moderate or severe asthma exacerbation less than 4 weeks prior to study entry.
* Subjects whose pharmacological therapy for asthma was modified in the 3 months prior to study entry.
* Subjects diagnosed with at least one of the following:

  * Lung cancer
  * Pulmonary fibrosis
  * Allergic bronchopulmonary aspergillosis
  * Eosinophilic granulomatosis with polyangiitis
  * Clinically relevant bronchiectasis or bronchiectasis associated with cystic fibrosis and/or allergic bronchopulmonary aspergillosis.
  * Chronic obstructive pulmonary disease associated with a smoking history ≥10 pack-years and/or history of exposure to biomass fuel combustion
* Subjects who are currently smokers or who have a history of smoking ≥ 10 pack-years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include adult patients with severe asthma, as per the definition of the International ERS/ATS Guidelines on Definition, Evaluation and Treatment of Severe Asthma, and who attend their routine clinical appointment at Brazilian centres specialized in the management of severe asthma.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of an eosinophilic phenotype of blood eosinophil count > 300 cells/mm3 among severe asthma patients in Brazil. | 8-month

SECONDARY OUTCOMES:
Prevalence of an eosinophilic phenotype of blood eosinophil count > 150 cells/mm3. | 8-month
Prevalence of an atopic phenotype, defined by a pre-existing history of atopy and total serum IgE > 100 UI/mL. | 8-month
Prevalence of atopy, as defined by a pre-existing history of atopy and total serum IgE > 100 UI/mL, among patients that present an eosinophilic phenotype of blood eosinophil count > 300 cells/mm3. | 8-month
Annual exacerbation rate. | 12-month
Patient-reported QoL using the St. George's Respiratory Questionnaire (SGRQ) results. | 8-month
  The SGRQ allows for the assessment of QoL of asthma patients. The questionnaire evaluates three domains: patient's perception of their recent respiratory problems (Symptoms score), disturbances to daily physical activity (Activity score) and disturbances of psycho-social function (Impact score). The score of each component and a total score can be computed. Scores are expressed as a percentage of overall impairment, where 100 represent the worst health status and 0 indicates the best status. Variables to collect: Symptoms score, Activity score, Impact score and Total score.
Asthma control using the Asthma Control Questionnaire 7 (ACQ 7) results. | 8-month
  The ACQ 7 allows for the evaluation of asthma control. Subjects will be asked to respond to six questions pertaining to asthma-related symptoms and bronchodilator use on a 7-point scale (where 0=no impairment and 6=maximum impairment). The seventh question will be answered by the study's team at the research center and involves scoring the FEV1% predicted on a 7-point scale. The total ACQ 7 score is computed through the mean of the 7 questions and, as such, varies between 0 (totally controlled asthma) and 6 (severely uncontrolled asthma). Variables to collect include the responses to each of the questionnaire's individual items.
Burden of disease using the GAD 7 scale. | 8-month
  The Generalized Anxiety Disorder (GAD -7) is a self-administered patient questionnaire used as a screening tool and as a severity measure for patients with generalized anxiety disorder. It is composed by 7 items: (1) feeling nervous, (2) not being able to stop or control worrying, (3) worrying too much about different things, (4) trouble relaxing, (5) being so restless that it is hard to sit still, (6) becoming easily annoyed or irritable, and (7) feeling afraid as if something awful might happen. Through a 4-point Likert scale from 'not at all' to 'nearly every day', it is asked how often the patient has been bothered by any of the presented problems. The GAD-7 index is obtained by adding the scores from the questionnaire, after having assigned 0 to the least severe situation, 3 to the most severe one, and 1 and 2 to the intermediate ones. The cut off points 5, 10 and 15 allow to classify the anxiety as none/normal (0-4), mild (5-9), moderate (10-14), and severe (15-21).
Burden of disease using the PHQ-9. | 8-month
  The Patient Health Questionnaire (PHQ) is a self-administered instrument for common mental disorders. The PHQ-9 is the depression module from the full PHQ and consists of 9 questions that assess the presence of each of the symptoms for the episode of major depression. The PHQ-9 score can range from 0-27, since each of the 9 items can be scored from 0-3 corresponding to "no at all", "several days", "more than half the days" and "nearly every day" responses, respectively. Major depression is diagnosed if 5 or more symptoms have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. Other depression is diagnosed if 2, 3, or 4 symptoms have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. One of the 9 symptom ("thoughts that you would be better off dead or of hurting yourself in some way") counts if present at all, regardless of duration.
Burden of disease using the WPAI: Asthma questionnaire results. | 8-month
  The WPAI assess the subject's ability to work and perform regular activities. The questionnaire inquiries about the number of days and hours missed from work or general activities. It also asks patients to rate, on a scale from 0 to 10, the degree to which asthma impairs productivity at work and their ability to perform normal daily activities. Higher values represent a more-severe impact. Variables to collect include the responses to each of the questionnaire's individual items.
Chronic oral corticosteroid (OCS) rate. | 8-month

CONTACTS AND LOCATIONS:
Overall Officials: Adelmir Machado, MD, Principal Investigator — Associação PROAR - Associação do Programa de Controle da Asma e da Rinite Alérgica na Bahia; Faradiba Serpa, MD, Principal Investigator — Santa Casa de Misericórdia de Vitória; Marcelo Rabahi, MD, Principal Investigator — CLARE - CLINICA DE PNEUMOLOGIA S/S; Daniela Blanco, MD, Principal Investigator — Hospital São Lucas da PUCRS; Marina Lima, MD, Principal Investigator — Hospital DIA do Pulmão / Complexo de Prevenção, Diagnóstico, Terapia e Reabilitação Respiratória LTDA; Rafael Stelmach, MD, Principal Investigator — InCor - Instituto do Coração - HCFMUSP.; Pedro Francisco Giovina-Bianchi Júnior, MD, Principal Investigator — HCUSP - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Alcindo Cerci Neto, MD, Principal Investigator — Universidade Estadual de Londrina; Martti Antila, MD, Principal Investigator — Clínica de Alergia Martti Antila / CMPC Pesquisa Clínica; Luisa Karla Arruda, MD, Principal Investigator — HCUSP RP - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo
Locations (6):
- Brazil (6):
  - Research Site, Blumenau
  - Research Site, Goiânia
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, São Paulo
  - Research Site, Sorocaba

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00045&attachmentIdentifier=01e2b893-e263-4990-81fc-be92f8cc31a0&fileName=2020-08-06_BRAEOS_CSR_Synopsis.pdf&versionIdentifier=